CLINICAL TRIAL: NCT02213185
Title: Effect of EMLA® Patches for Reducing Pain Associated With Sterile Water Injections - a Randomized Controlled Trial
Brief Title: EMLA and Sterile Water Injections - Pain From Injections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Skövde (Other)
Responsible Party: Principal Investigator, Lena B Martensson, Professor, University of Skövde
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: O-9-2013
Record Dates: First submitted 2014-08-07; First posted 2014-08-11 (Estimated); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Pain
Keywords: Sterile water injections; Pain; VAS; Complementary method
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- EMLA patches and SWI (Experimental): EMLA patches 1.5 hrs before sterile water injections
  Interventions: Other: EMLA patches
- EMLA patches and isotonic saline (Active Comparator): EMLA patches 1.5 hrs before isotonic saline
  Interventions: Other: EMLA patches
- Placebo patches and SWI (Placebo Comparator): PLACEBO patches 1.5 hrs before sterile water injections
  Interventions: Other: EMLA patches
- Placebo patches and isotonic saline (Placebo Comparator): PLACEBO patches 1.5 hrs before isotonic saline
  Interventions: Other: EMLA patches

INTERVENTIONS:
Other: EMLA patches — EMLA patches 1.5 hrs before sterile water injections

SUMMARY:
The aim is to study the effect of local anaesthesia (EMLA®) on pain associated with sterile water injections.

DETAILED DESCRIPTION:
Sterile Water Injection (SWI) was previously shown to give good pain relief for lower-back pain during childbirth, chronic neck pain and ureterolithiasis. However, the pain associated with the injections remains problematic, and therefore it is important to find a less painful injection technique.

ELIGIBILITY:
Inclusion Criteria

* Woman
* Age 18-45 years
* Healthy
* Ability to understand information and instructions

Exclusion Criteria:

* Pregnancy
* Previous experience of SWI
* On-going pain
* Use of medication for depression, pain, or sleeping disorder 24 hours prior to the experiment
* Smoking, snuffing, physical activity, and intake of caffeinated beverages (coffee, tea, or energy drink (e.g., Red Bull) 2 hours prior to the experiment

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2019-12-18 (Actual); Study Completion 2019-12-18 (Actual)

PRIMARY OUTCOMES:
Self reported experience of injection pain measured by Visual Analogue Scale following Sterile Water Injections | 15 minutes
  Self reported experiences of pain with Visual Analogue Scale 0=no pain 10=worst imaginable pain

SECONDARY OUTCOMES:
Self reported (questionnaire descriptive via email), self-reported experiences of side effects following Sterile Water injections | 24 hours
  Self reported (questionnaire descriptive via email), self-reported experiences of of side effects following Sterile Water injections

CONTACTS AND LOCATIONS:
Overall Officials: Lena B Mårtensson, Professor, Principal Investigator — University of Skövde
Locations (1):
- School of Health Sciences, University of Skövde, Skövde, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Martensson LB, Gunnarsson BM, Karlsson S, Lee N, Bergh I. Effect of topical local anaesthesia on injection pain associated with administration of sterile water injections - a randomized controlled trial. BMC Anesthesiol. 2022 Feb 1;22(1):35. doi: 10.1186/s12871-022-01573-0. PMID 35105307